CLINICAL TRIAL: NCT01716819
Title: Role of the Renin Angiotensin Aldosterone System and Remodeling of the Matrix Cardiac Extra Cellular in the Mechanisms of Transition to Heart Failure in Abdominal Obesity: Prospective Longitudinal Study R2C2 II
Brief Title: Role of the Renin Angiotensin Aldosterone System in the Mechanisms of Transition to Heart Failure in Abdominal Obesity
Acronym: R2C2-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-A00574-39
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Obesity, Abdominal
Keywords: Heart failure, abdominal obesity, RAAS
MeSH Terms: conditions — Obesity, Abdominal; Heart Failure | interventions — Blood Specimen Collection; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abdominal obesity (Other): Single arm, follow up cohort in patient with abdominal obesity. No comparator: description of interventions :
  Composition of body mass by Dual x-ray absorptiometry Pulse wave velocity Electrocardiogram Urine sample Blood sample (and biological collection) Assessment of sleep apnea syndrome Glucose tolerance test Echocardiography Echotracking cardiac and abdominal magnetic resonance imaging Ambulatory blood pressure monitoring
  Interventions: Other: Urine sample; Other: Blood sample; Other: Assessment of sleep apnea syndrome; Other: Electrocardiogram; Other: Glucose tolerance test; Other: Echocardiography; Other: cardiac and abdominal magnetic resonance imaging; Other: Ambulatory blood pressure monitoring; Other: Echotracking; Other: Pulse wave velocity; Other: Composition of body mass by Dual x-ray absorptiometry

INTERVENTIONS:
Other: Urine sample — dosages on one spot and 24h collection
Other: Blood sample — dosages
Other: Assessment of sleep apnea syndrome
Other: Electrocardiogram
Other: Glucose tolerance test
Other: Echocardiography
Other: cardiac and abdominal magnetic resonance imaging
Other: Ambulatory blood pressure monitoring
Other: Echotracking
Other: Pulse wave velocity
Other: Composition of body mass by Dual x-ray absorptiometry

SUMMARY:
R2C2 study has shown that abdominal obesity is associated with a cardiac and vascular remodelling in healthy volunteers. This remodelling is correlated with renin-angiotensin aldosterone system (RAAS) activation and/or systemic fibrosis. R2C2 II study is designed to confirm the hypothesis that RAAS is associated with an early remodelling and implicated in the transition to cardiac failure in abdominal obesity.

DETAILED DESCRIPTION:
Follow up of abdominal obesity patients from the R2C2 cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Being a former member of R2C2 study, abdominal obese group.
* Having signed the informed consent (refusing to participate to the genetic study is not an exclusion criteria).
* being affiliated to health insurance scheme.

Inclusion Criteria of R2C2 study:

* Men and women aged between 40 and 65 year's old
* Caucasian
* Born or living in France for at least 10 years
* Presenting an abdominal obesity defined by a waist circumference >94 cm in men and ≥ 80 cm in women, associated or not with untreated hypertension or hypertension treated for less than one year
* Having signed the informed consent

Exclusion Criteria:

* Subjects unable to understand the information letter
* Subjects under supervision or guardianship
* pregnant or lactating woman
* A contraindication to perform MRI is not an exclusion criteria.

Ages: 43 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
cardiac extracellular matrix remodelling | 3-7 years
  Initial values of cardiac extracellular matrix remodelling biomarkers and the evolution of biomarkers at 3-7 years

SECONDARY OUTCOMES:
Cardiac and arterial phenotype | 3-7 years
  Evolution of cardiac and vascular phenotype in 3-7 years.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick ROSSIGNOL, Principal Investigator — CIC-P - INSERM - Institut Lorrain du Cœur et des vaisseaux Louis Mathieu
Locations (1):
- CIC-P - INSERM - Institut Lorrain du Cœur et des vaisseaux, Vandœuvre-lès-Nancy, Meurthe et Moselle, France

REFERENCES:
- [Derived] Mandry D, Girerd N, Lamiral Z, Huttin O, Filippetti L, Micard E, Beaumont M, Ncho Mottoh MB, Pace N, Zannad F, Rossignol P, Marie PY. Relationship Between Left Ventricular Ejection Fraction Variation and Systemic Vascular Resistance: A Prospective Cardiovascular Magnetic Resonance Study. Front Cardiovasc Med. 2021 Dec 24;8:803567. doi: 10.3389/fcvm.2021.803567. eCollection 2021. PMID 35004914